CLINICAL TRIAL: NCT04478591
Title: The Wearing-off Phenomenon of Ocrelizumab in Patients With Multiple Sclerosis
Acronym: WOC
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Zoé van Kempen, principal investigator, Amsterdam UMC, location VUmc
Other Study IDs: 2020.191
Record Dates: First submitted 2020-06-24; First posted 2020-07-20 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Ocrelizumab; Wearing-off effect; Neurofilament Light; Extended dosing
MeSH Terms: conditions — Multiple Sclerosis; Charcot-Marie-Tooth disease, Type 1F | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with multiple sclerosis using ocrelizumab.: Patients with multiple sclerosis using ocrelizumab for a minimum of one year.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — All participants will fill in two questionnaires before or during their next treatment with ocrelizumab: the MSIS-29 questionnaire and a wearing-off questionnaire. After two weeks, participants fill in two digital questionnaires (MSIS-29, additional wearing-off questionnaire).

SUMMARY:
The primary goal of this research is to study the prevalence of the wearing-off effect and possible risk factors for wearing-off symptoms in patients with multiple sclerosis using ocrelizumab with the use of questionnaires. Furthermore, the goal is to study whether patients receiving extended dosing of ocrelizumab experience more wearing-off symptoms or adverse events in general. Finally, we would like to extend knowledge on wearing-off symptoms in general.

DETAILED DESCRIPTION:
Ocrelizumab is a monoclonal antibody very effective for the treatment of relapsing-remitting multiple sclerosis and primary progressive multiple sclerosis. Ocrelizumab is usually administered intravenous every six months. Natalizumab is another type of treatment used for relapsing-remitting multiple sclerosis and is administered every four weeks. Often patients report MS-related symptoms just prior to their next infusion such as fatigue, coordination problems or motor problems, the so-called wearing-off phenomenon. The exact etiology of this phenomenon remains unknown. Although not studied before, patients do report similar symptoms when using ocrelizumab. Furthermore, because of the COVID-19 pandemic, some patients receive extended dosing of ocrelizumab based on b-cell count. Whether this can increase wearing-off symptoms is unknown.

The goal of this research is to study the prevalence of wearing-off symptoms and possible risk factors for wearing-off symptoms in patients with multiple sclerosis using ocrelizumab. All patients using ocrelizumab during one year or more that provided written informed consent to participate in the study will be asked to complete three questionnaires before or during their next treatment with ocrelizumab. The questionnaires that will be used are the MSIS-29, the treatment satisfaction questionnaire and a questionnaire about wearing-off symptoms. Exact weight of the participants will be measured. Information about age, gender, date of diagnosis, start date of ocrelizumab, clinical and radiological disease activity, EDSS score, b-cell count and the biomarker neurofilament light will be extracted from the patient files. After two weeks, participants receive two additional digital questionnaires, the MSIS-29 and a follow-up questionnaire about wearing-off symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diagnosis multiple sclerosis
* Use of ocrelizumab as a treatment for multiple sclerosis for a minimum of one year

Exclusion Criteria:

* Unable to answer questionnaires in Dutch
* Different infusion protocol during the previous ocrelizumab infusion (e.g. 300 mg of ocrelizumab instead of 600 mg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multiple sclerosis using ocrelizumab.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Wearing-off symptoms | Baseline
  Prevalence of wearing-off symptoms prior to ocrelizumab infusion (yes/no assessed on questionnaires)

SECONDARY OUTCOMES:
% of wearing-off symptoms (yes/no assessed on questionnaires) in correlation to the % of patients with extended dosing versus standard dosing with ocrelizumab. | At baseline (prior to next infusion with ocrelizumab)
  % of wearing-off symptoms (yes/no assessed on questionnaires) in correlation to the % of patients with extended dosing versus standard dosing with ocrelizumab.
Neurofilament light levels in patients with wearing-off symptoms. | At baseline (prior to next infusion with ocrelizumab)
  Neurofilament light levels in patients with wearing-off symptoms compared to patients without wearing-off symptoms.
Absolute B-cells count in blood in correlation to the presence of wearing-off symptoms (yes/no assessed on questionnaires) | At baseline (prior to next infusion with ocrelizumab)
  Absolute B-cells count in blood in correlation to the presence of wearing-off symptoms (yes/no assessed on questionnaires) levels in patients with wearing-off symptoms.
Type of multiple sclerosis (either RRMS or PPMS) in correlation to % of patients with wearing-off symptoms (yes/no assessed on questionnaires). | At baseline (prior to next infusion with ocrelizumab)
  Type of multiple sclerosis (either RRMS or PPMS) in correlation to % of patients with wearing-off symptoms (yes/no assessed on questionnaires).
Treatment satisfaction score measured by the treatment satisfaction questionnaire in correlation to the % of patients with wearing-off symptoms (yes/no assessed on questionnaires) | At baseline (prior to next infusion with ocrelizumab)
  Treatment satisfaction score measured by the treatment satisfaction questionnaire in correlation to the % of patients with wearing-off symptoms (yes/no assessed on questionnaires)
Self-reported disability (MSIS-29 questionnaire) compared before and after ocrelizumab infusion in patients with wearing-off symptoms | At baseline (prior to next infusion with ocrelizumab) and after two weeks
  Self-reported disability before ocrelizumab infusion compared before and after ocrelizumab (delta scores) in patients with wearing-off symptoms
Self-reported disability (MSIS-29 questionnaire) after ocrelizumab infusion in patients without wearing-off symptoms | At baseline (prior to next infusion with ocrelizumab) and after two weeks
  Self-reported disability after ocrelizumab infusioSelf-reported disability before ocrelizumab infusion compared before and after ocrelizumab (delta scores) in patients with wearing-off symptomsn in patients without wearing-off symptoms
Change of wearing-off symptoms after ocrelizumab infusion in patients with wearing-off symptoms | Two weeks after ocrelizumab infusion
  Change of wearing-off symptoms after ocrelizumab infusion in patients with wearing-off symptoms as measured with the wearing-off questionnaire (questionnaire designed for this study evaluating wearing-off symptoms).
Post-dose symptoms after ocrelizumab infusion | Two weeks after ocrelizumab infusion
  Post-dose symptoms after ocrelizumab infusion as measured with the wearing-off questionnaire (questionnaire designed for this study evaluating wearing-off symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Joep Killestein, MD, PhD., Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Amsterdam UMC, location VUmc, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided